CLINICAL TRIAL: NCT00761839
Title: Does Use of a Wound After-care Summary Improve Patient Satisfaction and Time to Wound Healing?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was withdrawn because of a problem with the software used for generating the aftercare summary.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XVA 41-027
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Wounds
Keywords: wound healing; self-management; patient education
MeSH Terms: conditions — Wounds and Injuries | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): These patients receive the experimental intervention--the after-care summary.
  Interventions: Behavioral: After-care summary
- Arm 2 (Active Comparator): These patients are the control group and receive usual care.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: After-care summary — The wound care NP will measure the wound and assess adherence to the following self-management activities: visiting the wound care clinic as scheduled; offloading; applying dressings; obtaining assistance at home; and participating in social activities. This information will be entered into a computer database on a VA computer that will generate a summary chart showing the relationship between adherence and wound healing. The generated "after-care summary" will be discussed with the patient and used to set self-management goals.
  Arms: Arm 1
Behavioral: Control group — Patients in the control group will receive usual counseling for self-management.
  Arms: Arm 2

SUMMARY:
The purpose of this research study is to evaluate a patient education program for chronic wound care. The wound care nurse practitioner (NP) at the Ann Arbor VAMC will use a wound self-management "after-care summary" with approximately half of her patients. This study will examine whether using this patient education tool for self-management of wound care results in improved patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

All patients presenting for outpatient wound care at the Ann Arbor VA Medical Center NP wound care clinic, who meet the following inclusion criteria for chronic wounds: stage II, III, IV pressure ulcers; venous stasis ulcers, and diabetic ulcers.

Exclusion Criteria:

Cognitively impaired patients who cannot give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
patient satisfaction, frequency of self-management activities, time to healing | Outcomes are measured at each participating patient's visit for one year or until the patient's wound is healed, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Julie C Lowery, PhD MHSA, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington